CLINICAL TRIAL: NCT06138821
Title: Effect of Endoscopic Sleeve Gastroplasty on Patients With Obesity and Concomitant Metabolic Dysfunction-Associated Steatohepatitis (MASH): A Multicenter, Open-label, Randomized Controlled Trial
Brief Title: Effect of Endoscopic Sleeve Gastroplasty in Patients With Obesity and MASH: A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pichamol Jirapinyo, MD, MPH (Other)
Collaborators: Boston Scientific Corporation (Industry); Cook Group Incorporated (Industry)
Responsible Party: Sponsor-Investigator, Pichamol Jirapinyo, MD, MPH, Director of Bariatric Endoscopy Fellowship, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024P002282
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Liver Diseases; Liver Fibrosis; Liver Fat; Metabolic Dysfunction-Associated Steatotic Liver Disease; Metabolic Dysfunction-Associated Steatohepatitis; MASLD; MASH; Weight Loss; Insulin Resistance; Insulin Sensitivity; Insulin Sensitivity/Resistance; Metabolic Disease; Diabetes; Diabetes Mellitus, Type 2; NASH With Fibrosis; Non-Alcoholic Fatty Liver Disease; Non Alcoholic Fatty Liver; Non-alcoholic Steatohepatitis
Keywords: Gut Hormones; Endoscopic Bariatric and Metabolic Therapy (EBMT); Intragastric Balloon (IGB); Endoscopic Suturing; Endoscopic Sleeve Gastroplasty (ESG); Weight Management; Endoscopic Gastric Remodeling (EGR); Endoscopic Bariatric Therapy (EBT); Fatty Liver; Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD); Metabolic Dysfunction-Associated Steatohepatitis (MASH); Non-Alcoholic Fatty Liver Disease (NAFLD); Non-Alcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Obesity; Liver Diseases; Liver Cirrhosis; Fatty Liver; Weight Loss; Insulin Resistance; Metabolic Diseases; Diabetes Mellitus; Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: This study is a randomized, controlled, open-label clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ESG + lifestyle modification (Experimental): Endoscopic sleeve gastroplasty weight loss procedure with a lifestyle modification program for 12 months.
  Interventions: Device: ESG + lifestyle modification; Behavioral: Lifestyle modification
- Lifestyle modification (Active Comparator): Lifestyle modification program for 12 months.
  Interventions: Behavioral: Lifestyle modification

INTERVENTIONS:
Device: ESG + lifestyle modification — Endoscopic sleeve gastroplasty - an endoscopic weight loss procedure where an endoscopic suturing device is utilized to reduce the size of the stomach by 70%.
  Other Names: Endoscopic sleeve gastroplasty; Endoscopic suturing
  Arms: ESG + lifestyle modification
Behavioral: Lifestyle modification — Lifestyle modification program consisting of diet and exercise therapy

SUMMARY:
Metabolic dysfunction-associated steatotic liver disease (MASLD) is the most common chronic liver disease globally. While weight loss through lifestyle modification is the standard treatment, most patients regain weight limiting ultimate improvement in liver disease. On the other end of the spectrum, bariatric surgery has shown promise in the treatment of MASLD/metabolic dysfunction-associated steatohepatitis (MASH) due to its efficacy in inducing weight loss. Nevertheless, its adoption has been hindered by the perceived invasiveness of surgery.

Over the past decade, endoscopic sleeve gastroplasty (ESG) has gained recognition as a promising minimally-invasive approach to weight loss. The procedure involves utilizing a Food and Drug Administration (FDA)-authorized endoscopic suturing device to reduce the gastric volume by 70%. Studies reveal that ESG is associated with approximately 18.2% weight loss at one year after the procedure, with sustained results for at least 10 years. Nevertheless, the effect of ESG on MASH remains unknown.

In this study, the investigators will compare ESG + lifestyle modification versus lifestyle modification alone in treating histologic MASH. The study will randomize patients to one of two different treatment options: ESG + lifestyle modification or lifestyle modification alone.

DETAILED DESCRIPTION:
The National Institutes of Health, the World Health Organization, and numerous other scientific organizations including the America Medical Association (AMA) recognize obesity as a chronic disease requiring primary therapy. Almost half of United States (U.S.) adults have obesity. The increasing prevalence of obesity in the U.S. has been accompanied by an increasing prevalence in its associated comorbid conditions including hypertension, diabetes, dyslipidemia, coronary heart disease, stroke, sleep apnea, osteoarthritis, gallbladder disease, GERD, and metabolic dysfunction-associated steatotic liver disease (MASLD)/metabolic dysfunction-associated steatohepatitis (MASH). Obesity is associated with an increased risk of all-cause and cardiovascular mortality and accounts for about 2.5 million preventable deaths annually. The economic consequences of MASH are enormous, with the lifetime cost of care for all patients with MASH projected to be approximately $222 billion as of 2017.

Current treatment options for patients with MASLD/MASH are limited to weight loss via lifestyle modification and more recently, Food and Drug Administration (FDA)-approved medications, such as resmetirom and semaglutide, indicated specifically for patients with MASH and F2-F3 fibrosis. Nevertheless, less than 10% of patients who undergo lifestyle modification experience at least 10% total weight loss (TWL), the threshold required for hepatic fibrosis regression. The available pharmacological approaches for the treatment of obesity increase weight loss by 3% to 9% compared with lifestyle therapy alone, but some can be associated with unfavorable side effects, significant cost, and weight loss achieved by pharmacotherapy is rarely maintained upon withdrawal of the medication. On the other end of the spectrum, bariatric surgery, such as Roux-en-Y gastric bypass (RYGB) and sleeve gastrectomy, has shown promise in the treatment of MASLD/MASH due to its ability to induce significant and durable weight loss of at least 10% TWL. Nevertheless, its adoption has been limited with less than 2% of patients eligible for the surgery choosing to undergo the procedure. This is likely due to the perceived invasiveness of surgery, high costs, and limited access. More importantly, the majority of patients with mild to moderate (class I and class II obesity (BMI 30-40 kg/m2)), who do not qualify for bariatric surgery are left without an effective management, considering the modest effects seen with medications or lifestyle intervention alone and their ability to achieve >10%TWL only in the minority of patients. Yet, according to the global disability-adjusted life-years and deaths study, patients with mild to moderate obesity are the highest contributors to the burden on disease both in terms of co-morbidities and overall mortality. Therefore, both government agencies (the Agency for Healthcare Research and Quality [AHRQ]) and national societies (American Society of Bariatric and Metabolic Surgery [ASMBS], and American Society of Gastrointestinal Endoscopy [ASGE]) now recognize that a significant management gap exists for patients with mild to moderate obesity and have defined safety and efficacy thresholds for adoption of a new treatment category- endoscopic weight loss interventions.

Over the past decades, endoscopic bariatric and metabolic therapies (EBMTs) have been developed to fill the treatment gap for obesity and MASLD/MASH. Specifically, compared to lifestyle modification, EBMTs are associated with greater weight loss with a higher proportion of patients reaching the 10% TWL threshold. Additionally, given its non-surgical, minimally-invasive nature, the safety profile for EBMTs appears more favorable compared to bariatric surgery. To date, there are two EBMT devices and/or procedures that are approved or cleared by the Food and Drug Administration (FDA). These include intragastric balloons (IGBs) and endoscopic sleeve gastroplasty (ESG).

The ESG procedure is an endoscopic minimally-invasive weight loss procedure where a commercially available, FDA-approved, full-thickness endoscopic suturing device (Overstitch; Boston Scientific, Marlborough, MA) is used to reduce the stomach volume by 70% through the creation of a restrictive endoscopic sleeve. This is accomplished by a series of endoluminally placed full-thickness stitches through the gastric wall, extending from the distal gastric body to the proximal gastric body. The investigators currently perform this procedure as a standard of care at Brigham and Women's Hospital (BWH). Our previous studies have demonstrated that ESG not only leads to significant weight loss of at least 10% TWL, but also improves non-invasive tests (NITs) of liver steatosis and fibrosis, as well as MASH histologic features in patients with obesity and concomitant MASH. Nevertheless, it remains unclear if ESG is superior to lifestyle modification alone.

Clinical Data to Date

The feasibility of ESG was first demonstrated in humans in the US in 2013. Since then, the technique has gained wide clinical adoption in the US and worldwide with thousands of cases performed. Multiple single-arm prospective and retrospective studies have demonstrated the safety and minimally invasive nature of the technique and reported %TWL of about 16% to 18% at 12 months. Furthermore, studies have demonstrated physiologic perturbations resulting from creation of the ESG and its association with increased satiation and metabolic effects that are potentially important to control the metabolic dysregulation associated with obesity. In a recent randomized controlled trial including 209 participants, subjects were randomized to either ESG combined with lifestyle modification (n=85) or lifestyle modification alone (n=124). At 12 months, the ESG group achieved significantly greater weight loss of 13.6% TWL, compared to 0.8% in the control group. ESG-related serious adverse events occurred in only 2% of participants, with no instances of mortality, intensive care, or surgery required. While ESG has demonstrated both safety and efficacy for weight loss, no RCTs have yet assessed its impact on obesity-related comorbidities.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 (male or female)
2. BMI ≥30 kg/m2
3. Self-reported stable weight (no weight change >5%) for 6 months prior to the first study visit
4. Willingness to follow protocol requirements, including signed informed consent, routine follow-up schedule, completing laboratory/imaging/additional tests, and completing diet counseling
5. Willingness to NOT start a new anti-obesity medication for the following 12 months
6. Residing within a reasonable distance from the investigator's office and able to travel to the investigator to complete routine follow-up visits
7. Ability to give informed consent
8. Women of childbearing potential (i.e., not post-menopausal, nor surgically sterilized) must agree to use adequate birth control methods

Exclusion Criteria:

1. Known history of other chronic liver diseases (viral hepatitis, autoimmune hepatitis, drug-induced hepatitis, and genetic)
2. Treatment with vitamin E (at doses ≥800 IU/day), pioglitazone, obeticholic acid, or resmetirom <90 days before the first study visit
3. History of foregut or gastrointestinal (GI) surgery (except uncomplicated fundoplication, cholecystectomy or appendectomy)
4. Prior bariatric surgery
5. Prior endoscopic sleeve gastroplasty
6. Any inflammatory disease of the GI tract, including severe (LA Grade C or D) esophagitis, Barrett's esophagus with dysplasia, gastric ulceration, duodenal ulceration, cancer or specific inflammation such as Crohn's disease
7. Potential upper gastrointestinal bleeding conditions such as esophageal or gastric varices, congenital or acquired intestinal telangiectasis, or other congenital anomalies of the gastrointestinal tract such as atresias or stenoses
8. Severe gastroesophageal reflux disease (GERD)
9. A structural abnormality in the esophagus or pharynx, such as a stricture or diverticulum, that could impede passage of the endoscope.
10. Achalasia or any other severe esophageal motility disorder
11. Chronic abdominal pain
12. Gastroparesis or intractable constipation
13. Hepatic insufficiency or cirrhosis
14. Severe coagulopathy
15. Insulin-dependent diabetes (either type 1 or type 2) or a significant likelihood of requiring insulin treatment in the following 12 months or HgbA1C ≥ 10%
16. Patients on an anti-platelet agent, anticoagulant agent or chronic/routine use of NSAIDs
17. Patients on corticosteroids, immunosuppressants, or narcotics
18. Patients on an anti-seizure or anti-arrhythmic medication
19. Patients who are pregnant or breastfeeding
20. Excessive alcohol consumption (>20 g per day for women; >30 g per day for men)
21. Active smoking
22. History of poorly controlled hypertension, coronary artery disease, congestive heart failure, cardiac arrhythmia
23. History of respiratory diseases such as chronic obstructive pulmonary disease (COPD) requiring steroids, pneumonia, or cancer
24. History of autoimmune connective tissue disorder such as lupus, scleroderma or immunocompromised disease
25. History of active malignancy
26. History of genetic or hormonal causes for obesity, such as Prader Willi syndrome
27. History of endocrine disorders affecting weight, such as uncontrolled hypothyroidism
28. Eating disorders, including night eating syndrome, bulimia, binge eating disorder or compulsive overeating
29. Active psychological issues preventing participation in a lifestyle modification program as determined by a psychologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
MASH resolution without worsening of liver fibrosis at 12 months | Baseline, 12 months
  Comparison of endoscopic ultrasound (EUS)-guided liver biopsy results to assess MASH resolution at 12 months compared to baseline in the ESG + lifestyle modification (LM) group compared to LM alone group.

SECONDARY OUTCOMES:
An improvement of liver fibrosis by at least one stage without worsening of MASH at 12 months | Baseline, 12 months
  Comparison of endoscopic ultrasound (EUS)-guided liver biopsy results to assess an improvement of liver fibrosis at 12 months compared to baseline in the ESG + lifestyle modification (LM) group compared to LM alone group.
Change in liver stiffness on MRE at 12 months | Baseline, 12 months
  Comparison of liver stiffness measurement on magnetic resonance elastography (MRE) at 12 months compared to baseline in the ESG + lifestyle modification (LM) group compared to LM alone group.
Change in liver stiffness on VCTE at 12 months | Baseline, 12 months
  Comparison of liver stiffness measurement on vibration-controlled transient elastography (VCTE) at 12 months compared to baseline in the ESG + lifestyle modification (LM) group compared to LM alone group.
Change in liver fibrosis using NFS at 12 months | Baseline, 12 months
  Comparison of NAFLD fibrosis score (NFS) at 12 months compared to baseline in the ESG + lifestyle modification (LM) group compared to LM alone group.
Change in liver fibrosis using ELF score at 12 months | Baseline, 12 months
  Comparison of ELF at 12 months compared to baseline in the ESG + lifestyle modification (LM) group compared to LM alone group.
Change in liver fibrosis using FIB-4 at 12 months | Baseline, 12 months
  Comparison of Fibrosis-4 (FIB-4) score at 12 months compared to baseline in the ESG + lifestyle modification (LM) group compared to LM alone group.
Change in liver fat content using MRI-PDFF at 12 months | Baseline, 12 months
  Comparison of liver fat content using MRI proton density fat fraction (MRI-PDFF) at 12 months compared to baseline in the ESG + lifestyle modification (LM) group compared to LM alone group.
Change in liver fat content using VCTE CAP score at 12 months | Baseline, 12 months
  Comparison of liver fat content measured by controlled attenuation parameter (CAP) score on vibration-controlled transient elastography (VCTE) at 12 months compared to baseline in the ESG + lifestyle modification (LM) group compared to LM alone group.
Change in portosystemic pressure gradient (PPG) measurements at 12 months | Baseline, 12 months
  Comparison of portosystemic pressure gradient (PPG) measurements at 12 months compared to baseline in the ESG + lifestyle modification (LM) group compared to LM alone group.
Percent total weight loss (%TWL) at 12 months | Baseline, 1, 3, 6 and 12 months
  Comparison of weight loss at 12 months compared to baseline in the ESG + lifestyle modification (LM) group compared to LM alone group.
Change in quality of life at 12 months | Baseline, 6 and 12 months
  Compare changes in quality of life assessed using chronic liver disease questionnaire at 12 months compared to baseline in the ESG + lifestyle modification (LM) group compared to LM alone group
Change in eating behaviors at 12 months | Baseline, 6 and 12 months
  Compare changes in eating behaviors evaluated using the Three Factor Eating Questionnaire (TFEQ) at 12 months compared to baseline in the ESG + lifestyle modification (LM) group compared to LM alone group.
Change in physical, mental and social well-being at 12 months | Baseline, 6 and 12 months
  Compare changes in physical, mental and social well-being using the Patient-reported Outcomes Measurement Information System (PROMIS) at 12 months compared to baseline in the ESG + lifestyle modification (LM) group compared to LM alone group.
Change in insulin resistance at 12 months | Baseline, 12 months.
  Compare changes in insulin resistance using Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) and Hemoglobin (HbA1c) values at 12 months compared to baseline in the ESG + lifestyle modification (LM) group compraed to LM alone group. groups
Change in gut hormones at 12 months | Baseline, 12 months.
  Compare changes in gut hormones using ghrelin, GIP, GLP-1, PYY values at 12 months compared to baseline in the ESG + lifestyle modification (LM) group compraed to LM alone group. groups
Change in bile acids at 12 months | Baseline, 12 months.
  Compare changes in bile acid values from blood samples at 12 months compared to baseline in the ESG + lifestyle modification (LM) group compraed to LM alone group. groups
Safety parameters post-procedure | Procedure day, 1, 3, 6, 9 and 12 months
  Rate of serious adverse events, defined as those classified as grade III-V according to the Clavien-Dindo classification in the ESG + LM group and LM alone group.

CONTACTS AND LOCATIONS:
Overall Officials: Pichamol Jirapinyo, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
De-identified data sharing will be considered on a case by case basis with a presentation of research protocol to the PI. Data will only be shared with a proper data transfer agreement in place between Brigham and Women's Hospital and the Institution of the requesting investigator.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 12 months after publication of study results. No end date.
Access Criteria: Data will only be shared with a proper data transfer agreement in place between Brigham and Women's Hospital and the Institution of the requesting investigator.

REFERENCES:
- [Background] Flegal KM, Carroll MD, Ogden CL, Curtin LR. Prevalence and trends in obesity among US adults, 1999-2008. JAMA. 2010 Jan 20;303(3):235-41. doi: 10.1001/jama.2009.2014. Epub 2010 Jan 13. PMID 20071471
- [Background] Flegal KM, Kit BK, Orpana H, Graubard BI. Association of all-cause mortality with overweight and obesity using standard body mass index categories: a systematic review and meta-analysis. JAMA. 2013 Jan 2;309(1):71-82. doi: 10.1001/jama.2012.113905. PMID 23280227
- [Background] Adams KF, Schatzkin A, Harris TB, Kipnis V, Mouw T, Ballard-Barbash R, Hollenbeck A, Leitzmann MF. Overweight, obesity, and mortality in a large prospective cohort of persons 50 to 71 years old. N Engl J Med. 2006 Aug 24;355(8):763-78. doi: 10.1056/NEJMoa055643. Epub 2006 Aug 22. PMID 16926275
- [Background] Prospective Studies Collaboration; Whitlock G, Lewington S, Sherliker P, Clarke R, Emberson J, Halsey J, Qizilbash N, Collins R, Peto R. Body-mass index and cause-specific mortality in 900 000 adults: collaborative analyses of 57 prospective studies. Lancet. 2009 Mar 28;373(9669):1083-96. doi: 10.1016/S0140-6736(09)60318-4. Epub 2009 Mar 18. PMID 19299006
- [Background] Finkelstein EA, Trogdon JG, Cohen JW, Dietz W. Annual medical spending attributable to obesity: payer-and service-specific estimates. Health Aff (Millwood). 2009 Sep-Oct;28(5):w822-31. doi: 10.1377/hlthaff.28.5.w822. Epub 2009 Jul 27. PMID 19635784
- [Background] Cawley J, Meyerhoefer C. The medical care costs of obesity: an instrumental variables approach. J Health Econ. 2012 Jan;31(1):219-30. doi: 10.1016/j.jhealeco.2011.10.003. Epub 2011 Oct 20. PMID 22094013
- [Background] Jensen MD, Ryan DH, Apovian CM, Ard JD, Comuzzie AG, Donato KA, Hu FB, Hubbard VS, Jakicic JM, Kushner RF, Loria CM, Millen BE, Nonas CA, Pi-Sunyer FX, Stevens J, Stevens VJ, Wadden TA, Wolfe BM, Yanovski SZ; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Obesity Society. 2013 AHA/ACC/TOS guideline for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2985-3023. doi: 10.1016/j.jacc.2013.11.004. Epub 2013 Nov 12. No abstract available. PMID 24239920
- [Background] Stevens VJ, Obarzanek E, Cook NR, Lee IM, Appel LJ, Smith West D, Milas NC, Mattfeldt-Beman M, Belden L, Bragg C, Millstone M, Raczynski J, Brewer A, Singh B, Cohen J; Trials for the Hypertension Prevention Research Group. Long-term weight loss and changes in blood pressure: results of the Trials of Hypertension Prevention, phase II. Ann Intern Med. 2001 Jan 2;134(1):1-11. doi: 10.7326/0003-4819-134-1-200101020-00007. PMID 11187414
- [Background] Gregg EW, Chen H, Wagenknecht LE, Clark JM, Delahanty LM, Bantle J, Pownall HJ, Johnson KC, Safford MM, Kitabchi AE, Pi-Sunyer FX, Wing RR, Bertoni AG; Look AHEAD Research Group. Association of an intensive lifestyle intervention with remission of type 2 diabetes. JAMA. 2012 Dec 19;308(23):2489-96. doi: 10.1001/jama.2012.67929. PMID 23288372
- [Background] Look AHEAD Research Group; Pi-Sunyer X, Blackburn G, Brancati FL, Bray GA, Bright R, Clark JM, Curtis JM, Espeland MA, Foreyt JP, Graves K, Haffner SM, Harrison B, Hill JO, Horton ES, Jakicic J, Jeffery RW, Johnson KC, Kahn S, Kelley DE, Kitabchi AE, Knowler WC, Lewis CE, Maschak-Carey BJ, Montgomery B, Nathan DM, Patricio J, Peters A, Redmon JB, Reeves RS, Ryan DH, Safford M, Van Dorsten B, Wadden TA, Wagenknecht L, Wesche-Thobaben J, Wing RR, Yanovski SZ. Reduction in weight and cardiovascular disease risk factors in individuals with type 2 diabetes: one-year results of the look AHEAD trial. Diabetes Care. 2007 Jun;30(6):1374-83. doi: 10.2337/dc07-0048. Epub 2007 Mar 15. PMID 17363746
- [Background] Yanovski SZ, Yanovski JA. Long-term drug treatment for obesity: a systematic and clinical review. JAMA. 2014 Jan 1;311(1):74-86. doi: 10.1001/jama.2013.281361. PMID 24231879
- [Background] Wing RR, Lang W, Wadden TA, Safford M, Knowler WC, Bertoni AG, Hill JO, Brancati FL, Peters A, Wagenknecht L; Look AHEAD Research Group. Benefits of modest weight loss in improving cardiovascular risk factors in overweight and obese individuals with type 2 diabetes. Diabetes Care. 2011 Jul;34(7):1481-6. doi: 10.2337/dc10-2415. Epub 2011 May 18. PMID 21593294
- [Background] Buchwald H, Oien DM. Metabolic/bariatric surgery worldwide 2011. Obes Surg. 2013 Apr;23(4):427-36. doi: 10.1007/s11695-012-0864-0. PMID 23338049
- [Background] GBD 2015 Obesity Collaborators; Afshin A, Forouzanfar MH, Reitsma MB, Sur P, Estep K, Lee A, Marczak L, Mokdad AH, Moradi-Lakeh M, Naghavi M, Salama JS, Vos T, Abate KH, Abbafati C, Ahmed MB, Al-Aly Z, Alkerwi A, Al-Raddadi R, Amare AT, Amberbir A, Amegah AK, Amini E, Amrock SM, Anjana RM, Arnlov J, Asayesh H, Banerjee A, Barac A, Baye E, Bennett DA, Beyene AS, Biadgilign S, Biryukov S, Bjertness E, Boneya DJ, Campos-Nonato I, Carrero JJ, Cecilio P, Cercy K, Ciobanu LG, Cornaby L, Damtew SA, Dandona L, Dandona R, Dharmaratne SD, Duncan BB, Eshrati B, Esteghamati A, Feigin VL, Fernandes JC, Furst T, Gebrehiwot TT, Gold A, Gona PN, Goto A, Habtewold TD, Hadush KT, Hafezi-Nejad N, Hay SI, Horino M, Islami F, Kamal R, Kasaeian A, Katikireddi SV, Kengne AP, Kesavachandran CN, Khader YS, Khang YH, Khubchandani J, Kim D, Kim YJ, Kinfu Y, Kosen S, Ku T, Defo BK, Kumar GA, Larson HJ, Leinsalu M, Liang X, Lim SS, Liu P, Lopez AD, Lozano R, Majeed A, Malekzadeh R, Malta DC, Mazidi M, McAlinden C, McGarvey ST, Mengistu DT, Mensah GA, Mensink GBM, Mezgebe HB, Mirrakhimov EM, Mueller UO, Noubiap JJ, Obermeyer CM, Ogbo FA, Owolabi MO, Patton GC, Pourmalek F, Qorbani M, Rafay A, Rai RK, Ranabhat CL, Reinig N, Safiri S, Salomon JA, Sanabria JR, Santos IS, Sartorius B, Sawhney M, Schmidhuber J, Schutte AE, Schmidt MI, Sepanlou SG, Shamsizadeh M, Sheikhbahaei S, Shin MJ, Shiri R, Shiue I, Roba HS, Silva DAS, Silverberg JI, Singh JA, Stranges S, Swaminathan S, Tabares-Seisdedos R, Tadese F, Tedla BA, Tegegne BS, Terkawi AS, Thakur JS, Tonelli M, Topor-Madry R, Tyrovolas S, Ukwaja KN, Uthman OA, Vaezghasemi M, Vasankari T, Vlassov VV, Vollset SE, Weiderpass E, Werdecker A, Wesana J, Westerman R, Yano Y, Yonemoto N, Yonga G, Zaidi Z, Zenebe ZM, Zipkin B, Murray CJL. Health Effects of Overweight and Obesity in 195 Countries over 25 Years. N Engl J Med. 2017 Jul 6;377(1):13-27. doi: 10.1056/NEJMoa1614362. Epub 2017 Jun 12. PMID 28604169
- [Background] ASGE Bariatric Endoscopy Task Force; Sullivan S, Kumar N, Edmundowicz SA, Abu Dayyeh BK, Jonnalagadda SS, Larsen M, Thompson CC. ASGE position statement on endoscopic bariatric therapies in clinical practice. Gastrointest Endosc. 2015 Nov;82(5):767-72. doi: 10.1016/j.gie.2015.06.038. Epub 2015 Aug 15. No abstract available. PMID 26282949
- [Background] Mahapatra MK, Karuppasamy M, Sahoo BM. Therapeutic Potential of Semaglutide, a Newer GLP-1 Receptor Agonist, in Abating Obesity, Non-Alcoholic Steatohepatitis and Neurodegenerative diseases: A Narrative Review. Pharm Res. 2022 Jun;39(6):1233-1248. doi: 10.1007/s11095-022-03302-1. Epub 2022 Jun 1. PMID 35650449
- [Background] Abu Dayyeh BK, Rajan E, Gostout CJ. Endoscopic sleeve gastroplasty: a potential endoscopic alternative to surgical sleeve gastrectomy for treatment of obesity. Gastrointest Endosc. 2013 Sep;78(3):530-5. doi: 10.1016/j.gie.2013.04.197. Epub 2013 May 24. PMID 23711556
- [Background] Sharaiha RZ, Kedia P, Kumta N, DeFilippis EM, Gaidhane M, Shukla A, Aronne LJ, Kahaleh M. Initial experience with endoscopic sleeve gastroplasty: technical success and reproducibility in the bariatric population. Endoscopy. 2015 Feb;47(2):164-6. doi: 10.1055/s-0034-1390773. Epub 2014 Nov 7. PMID 25380510
- [Background] Lopez-Nava G, Galvao MP, da Bautista-Castano I, Jimenez A, De Grado T, Fernandez-Corbelle JP. Endoscopic sleeve gastroplasty for the treatment of obesity. Endoscopy. 2015 May;47(5):449-52. doi: 10.1055/s-0034-1390766. Epub 2014 Nov 7. PMID 25380508
- [Background] Abu Dayyeh BK, Acosta A, Camilleri M, Mundi MS, Rajan E, Topazian MD, Gostout CJ. Endoscopic Sleeve Gastroplasty Alters Gastric Physiology and Induces Loss of Body Weight in Obese Individuals. Clin Gastroenterol Hepatol. 2017 Jan;15(1):37-43.e1. doi: 10.1016/j.cgh.2015.12.030. Epub 2015 Dec 31. PMID 26748219
- [Background] ASGE/ASMBS Task Force on Endoscopic Bariatric Therapy; Ginsberg GG, Chand B, Cote GA, Dallal RM, Edmundowicz SA, Nguyen NT, Pryor A, Thompson CC. A pathway to endoscopic bariatric therapies. Gastrointest Endosc. 2011 Nov;74(5):943-53. doi: 10.1016/j.gie.2011.08.053. No abstract available. PMID 22032311
- [Background] Mechanick JI, Youdim A, Jones DB, Timothy Garvey W, Hurley DL, Molly McMahon M, Heinberg LJ, Kushner R, Adams TD, Shikora S, Dixon JB, Brethauer S. Clinical practice guidelines for the perioperative nutritional, metabolic, and nonsurgical support of the bariatric surgery patient--2013 update: cosponsored by American Association of Clinical Endocrinologists, the Obesity Society, and American Society for Metabolic & Bariatric Surgery. Surg Obes Relat Dis. 2013 Mar-Apr;9(2):159-91. doi: 10.1016/j.soard.2012.12.010. Epub 2013 Jan 19. PMID 23537696
- [Background] Abu Dayyeh BK, Bazerbachi F, Vargas EJ, Sharaiha RZ, Thompson CC, Thaemert BC, Teixeira AF, Chapman CG, Kumbhari V, Ujiki MB, Ahrens J, Day C; MERIT Study Group; Galvao Neto M, Zundel N, Wilson EB. Endoscopic sleeve gastroplasty for treatment of class 1 and 2 obesity (MERIT): a prospective, multicentre, randomised trial. Lancet. 2022 Aug 6;400(10350):441-451. doi: 10.1016/S0140-6736(22)01280-6. Epub 2022 Jul 28. PMID 35908555
- [Background] Vilar-Gomez E, Martinez-Perez Y, Calzadilla-Bertot L, Torres-Gonzalez A, Gra-Oramas B, Gonzalez-Fabian L, Friedman SL, Diago M, Romero-Gomez M. Weight Loss Through Lifestyle Modification Significantly Reduces Features of Nonalcoholic Steatohepatitis. Gastroenterology. 2015 Aug;149(2):367-78.e5; quiz e14-5. doi: 10.1053/j.gastro.2015.04.005. Epub 2015 Apr 10. PMID 25865049
- [Background] Harrison SA, Bedossa P, Guy CD, Schattenberg JM, Loomba R, Taub R, Labriola D, Moussa SE, Neff GW, Rinella ME, Anstee QM, Abdelmalek MF, Younossi Z, Baum SJ, Francque S, Charlton MR, Newsome PN, Lanthier N, Schiefke I, Mangia A, Pericas JM, Patil R, Sanyal AJ, Noureddin M, Bansal MB, Alkhouri N, Castera L, Rudraraju M, Ratziu V; MAESTRO-NASH Investigators. A Phase 3, Randomized, Controlled Trial of Resmetirom in NASH with Liver Fibrosis. N Engl J Med. 2024 Feb 8;390(6):497-509. doi: 10.1056/NEJMoa2309000. PMID 38324483
- [Background] Jirapinyo P, Zucker SD, Thompson CC. Regression of Hepatic Fibrosis After Endoscopic Gastric Plication in Nonalcoholic Fatty Liver Disease. Am J Gastroenterol. 2023 Jun 1;118(6):983-990. doi: 10.14309/ajg.0000000000002087. Epub 2022 Dec 23. PMID 36597405
- [Background] Jirapinyo P, Thompson CC, Garcia-Tsao G, Zucker SD, Ryou M. The effect of endoscopic gastric plication on portosystemic pressure gradient in patients with nonalcoholic fatty liver disease and compensated advanced chronic liver disease. Endoscopy. 2024 Jan;56(1):56-62. doi: 10.1055/a-2146-8857. Epub 2023 Aug 2. PMID 37532114
- [Background] Jirapinyo P, Hadefi A, Thompson CC, Patai AV, Pannala R, Goelder SK, Kushnir V, Barthet M, Apovian CM, Boskoski I, Chapman CG, Davidson P, Donatelli G, Kumbhari V, Hayee B, Esker J, Hucl T, Pryor AD, Maselli R, Schulman AR, Pattou F, Zelber-Sagi S, Bain PA, Durieux V, Triantafyllou K, Thosani N, Huberty V, Sullivan S. American Society for Gastrointestinal Endoscopy-European Society of Gastrointestinal Endoscopy guideline on primary endoscopic bariatric and metabolic therapies for adults with obesity. Gastrointest Endosc. 2024 Jun;99(6):867-885.e64. doi: 10.1016/j.gie.2023.12.004. Epub 2024 Apr 19. PMID 38639680